CLINICAL TRIAL: NCT06035237
Title: The Effect of Cold Spray Applied Before Local Anaesthesia on Pain and Anxiety in Coronary Angiography Procedure: a Randomised Controlled Study
Brief Title: The Effect of Cold Spray Applied Before Local Anaesthesia
Acronym: EffectofCold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozkan Sir (Other)
Responsible Party: Sponsor-Investigator, Ozkan Sir, PhD student, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Özkan
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pain; Anxiety; Coronary Artery Disease
Keywords: Pain, anxiety, cold spray, angiography
MeSH Terms: conditions — Pain; Anxiety Disorders; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients in the experimental group were informed that cold spray would be applied to their arm in a supine position to reduce procedure-related pain. For femoral artery angiography, the central part of the inguinal access area was targeted, and for radial angiography, 2 cm above the styloid process of the radial bone was targeted, and cold spray (Chloroethyl spray) was applied for approximately 3 seconds from a height of 10 cm.
  Interventions: Other: Cold Spray
- Control Group (No Intervention): Pain levels recorded with the VAS were evaluated for patients after the procedure using the state anxiety scale. Pain levels for control group patients were also assessed and recorded within the sheath after intravenous solutions were given. Anxiety levels were recorded after the procedure was completed.

INTERVENTIONS:
Other: Cold Spray — Cold Spray: Cold sprays, composed of liquefied gases under high pressure, rapidly evaporate from the applied area, causing a sudden drop in skin temperature. This condition leads to the temporary desensitization of pain receptors or the activation of ion channels, resulting in the brief alleviation of pain sensation. Various medical, non-medical, and surgical methods are employed to manage pain. Cold sprays are among non-medical methods, including massage, cold application, and distraction techniques. Therefore, cold sprays cannot be prescribed like medication. They are used for local anesthesia in cases of acute trauma, injections, blood collection, vein puncture, and similar situations.
  Arms: Experimental Group

SUMMARY:
Coronary angiography is a reliable and valid method used in the diagnosis of Coronary Artery Disease (CAD). Coronary angiography is defined as the process of obtaining cineangiographic images by administering radio-opaque material to the coronary vessels via arterial route. Coronary angiography is frequently performed from brachial, radial and femoral arteries. The aim of coronary angiography is to determine the presence, localisation and extent of cardiovascular lesions.

Invasive interventions cause anxiety and pain in the patient, increase the level of anxiety and cause a number of negative effects such as increased use of sedative drugs, development of post-procedure complications, prolongation of the recovery process and hospitalisation time. It is stated that there is a positive relationship between reducing the anxiety of the patients and meeting the needs of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and above.
* Not having used any anesthetic substance before the procedure.
* Not having undergone angiography before.
* Having no communication problems.

Exclusion Criteria:

* Having previously undergone angiography.
* Having taken analgesics before angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Pain levels recorded with the Visual Analog Scale | 1 minute
  VAS was used to evaluate the pain of the patients. The scale consists of emotion adjectives in which each emotion experienced by the person at that moment is marked with a vertical line on a plane. A value of zero is considered as not experiencing pain at all, and a value of ten is considered as experiencing pain completely.

CONTACTS AND LOCATIONS:
Locations (1):
- Van yüzüncü yıl university, Van, Van, Turkey (Türkiye)